CLINICAL TRIAL: NCT01860547
Title: The Effect of the Bioactives of Sea Buckthorn and Bilberry on the Risk of Metabolic Diseases
Brief Title: Effects of Berries and Berry Fractions on Metabolic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Pakkasmarja (Other); Saarioinen (Other); Kiantama Ltd. (Unknown); Aromtech Ltd. (Industry); Fazer (Other); Satakunta Sea Buckthorn Society (Unknown); Finnish Berry Powders Ltd. (Unknown)
Responsible Party: Principal Investigator, Jukka-Pekka Suomela, University Lecturer, University of Turku
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TYBID1
Record Dates: First submitted 2013-04-29; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Type 2 Diabetes; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Vaccinium myrtillus extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- bilberry (Experimental)
  Interventions: Dietary Supplement: Bilberries
- sea buckthorn berry (Experimental)
  Interventions: Dietary Supplement: Sea buckthorn berry
- sea buckthorn phenolic extract (Experimental)
  Interventions: Dietary Supplement: Sea buckthorn phenolic extract
- sea buckthorn oil (Experimental)
  Interventions: Dietary Supplement: Sea buckthorn oil

INTERVENTIONS:
Dietary Supplement: Bilberries — Frozen bilberries, 100 g/d
  Arms: bilberry
Dietary Supplement: Sea buckthorn berry — Dried sea buckthorn berries, 20 g/d
  Arms: sea buckthorn berry
Dietary Supplement: Sea buckthorn phenolic extract — Ethanol-water extract from sea buckthorn berries, combined with maltodextrin, 14.6 g/d (7.3 g sea buckthorn extract + 7.3 g maltodextrin)
  Arms: sea buckthorn phenolic extract
Dietary Supplement: Sea buckthorn oil — Sea buckthorn oil, 4 g (8 capsules)/d
  Arms: sea buckthorn oil

SUMMARY:
The study hypothesis is that the bioactive compounds of sea buckthorn berries (Hippophaë rhamnoides), their fractions, and bilberries (Vaccinium myrtillus). have positive effects on lipid and carbohydrate metabolism and will thus reduce the risk of developing metabolic diseases.

DETAILED DESCRIPTION:
The aim of the project was to investigate whether it is possible to reduce the risk of metabolic diseases with supplementing the diet with sea buckthorn berries (Hippophaë rhamnoides), their bioactive fractions, and bilberries (Vaccinium myrtillus). The study design was a randomized cross-over clinical trial. The participants were slightly and moderately overweight female subjects. In total, 110 female volunteers were recruited, and they followed four different berry diets (bilberry, sea buckthorn, sea buckthorn phenolic extract and sea buckthorn oil) in a randomized order for 33-35 days. Each intervention was followed by a wash-out period of 30-39 days. Blood samples were drawn and physical measurements were performed after each period. Eighty volunteers completed the study. Different markers of lipid and carbohydrate metabolism and inflammation were measured form the blood samples.

ELIGIBILITY:
Inclusion Criteria:

* BMI 26-34
* total cholesterol 4.5-8 mmol/l
* LDL chol >2.5 mmol/l
* triglycerides <4 mmol/l
* glucose <6 mmol/l
* insulin <25 mU/l
* blood pressure <160/99 mm Hg
* hemoglobin >120 g/l
* thyroid-stimulating hormone 0.3-4.2 mU/l
* ALAT <60 U/l
* creatinine <115 umol/l

Exclusion Criteria:

* pregnancy
* menopause,
* regular smoking
* previously diagnosed diabetes (other than gestational)
* thyroid, renal, hematological, or hepatic dysfunction
* previous myocardial infarction
* cardiovascular medication
* treatment with regular medication other than allergy medication or joint lubricates
* on-going inflammatory disease

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Serum Alanine aminotransferase (ALAT) | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)

SECONDARY OUTCOMES:
Serum total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triacylglycerols | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Plasma glucose | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum gamma-glutamyl transpeptidase | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum high-sensitivity C-reactive protein | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum insulin | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum soluble intercellular adhesion molecule | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum tumor necrosis factor -alpha | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Body mass index | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum soluble vascular cell adhesion molecule | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum adiponectin | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Serum interleukine-6 | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Weight | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Waist circumference | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)
Body composition | Change from beginnig to end of each berry treatment (duration of treatments average 33-35 days)

OTHER OUTCOMES:
Subclasses of serum lipoproteins, serum fatty acids and lipid classes of serum | Change from beginning to end of each berry treatment (duration of treatments average 33-35 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jukka-Pekka Suomela, Ph.D., Principal Investigator — University of Turku; Heikki Kallio, Prof., Study Director — University of Turku
Locations (1):
- University of Turku, Dept of Biochemistry and Food Chemistry, Turku, Finland

REFERENCES:
- [Result] Lehtonen HM, Suomela JP, Tahvonen R, Yang B, Venojarvi M, Viikari J, Kallio H. Different berries and berry fractions have various but slightly positive effects on the associated variables of metabolic diseases on overweight and obese women. Eur J Clin Nutr. 2011 Mar;65(3):394-401. doi: 10.1038/ejcn.2010.268. Epub 2011 Jan 12. PMID 21224867
- [Derived] Larmo PS, Kangas AJ, Soininen P, Lehtonen HM, Suomela JP, Yang B, Viikari J, Ala-Korpela M, Kallio HP. Effects of sea buckthorn and bilberry on serum metabolites differ according to baseline metabolic profiles in overweight women: a randomized crossover trial. Am J Clin Nutr. 2013 Oct;98(4):941-51. doi: 10.3945/ajcn.113.060590. Epub 2013 Aug 14. PMID 23945716